CLINICAL TRIAL: NCT05191381
Title: Immune Modulation by Stem Cell Derived Exosomes in Critically Ill COVID-19
Brief Title: Immune Modulation by Exosomes in COVID-19
Acronym: IMECOV19
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, MBA, Clinical Professor, University of Ulm
Other Study IDs: Lung fibrosis in COVID19
Record Dates: First submitted 2022-01-12; First posted 2022-01-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Critical Illness; Hypercytokinemia; Lung Fibrosis
Keywords: COVID-19; Critical illness; Hypercytokinemia; Exosomes; Mesenchymal stem cells; Tissue reconstitution; Immune modulation; Sepsis
MeSH Terms: conditions — COVID-19; Critical Illness; Cytokine Release Syndrome; Pulmonary Fibrosis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — 4 ml of heparin- and 2 ml of EDTA-anti-coagulated blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: Application of exosomes in a whole blood assay — Co-incubation of patient-derived whole blood samples with mesenchymal stem cell derived exosomes and read-out of biomarkers, RNA and immune phenotypes after 24h.

SUMMARY:
Following whole blood stimulation with mesenchymal stem cell derived exosomes, immune phenotype, cytokine release and mRNA expression patterns from critically ill patients with COVID-19 will be determined.

DETAILED DESCRIPTION:
Critically ill patients with COVID-19 may develop lung failure and require extracorporal oxygenation due to hyperinflammation and progressive lung fibrosis. The anti-inflammatory and immune modulatory function of mesenchymal stem cells will be investigated by whole blood stimulation experiments using stem cell derived exosomes. Exosome preparations have been characterized by miRNA and protein expression patterns and suggest their tissue regenerative capacity.

The hypothesis of the present study is that mesenchymal stem cell derived exosomes attenuate inflammation and support anti-fibrotic pathways.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill COVID-19 patients with lung dysfunction
* COVID-19 WHO severity degree >= 4, ARDS (WHO Definition 13 March 2020)
* Body weight > 50 kg
* Informed consent

Exclusion Criteria:

* Pregnant or breast feeding women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill COVID-19 patients, COVID-19 WHO severity degree >= 4, ARDS (WHO Definition 13 March 2020)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine profile in supernatants | 24 hours, 1 year
  Quantification of pro- and anti-inflammatory biomarkers after 24 hours of whole blood culture

SECONDARY OUTCOMES:
Immune phenotyping | 1 year
  Immune phenotypes related to type I interferon signaling
Genetic predisposition to hyperinflammation | 1 year
  Determination of functional single nucleotide polymorphisms of inflammatory genes and receptors

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, Principal Investigator — Clinic of Anaesthesiology and Intensive Care Medicine; Marion Schneider, PhD, Principal Investigator — Clinic of Anaesthesiology and Intensive Care Medicine
Locations (1):
- Ulm University Hospital, Clinic of Anesthesiology and Intensive Care Medicine, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Di Rocco G, Baldari S, Toietta G. Towards Therapeutic Delivery of Extracellular Vesicles: Strategies for In Vivo Tracking and Biodistribution Analysis. Stem Cells Int. 2016;2016:5029619. doi: 10.1155/2016/5029619. Epub 2016 Nov 23. PMID 27994623
- [Background] Geistlinger J, Du W, Groll J, Liu F, Hoegel J, Foehr KJ, Pasquarelli A, Schneider EM. P2RX7 genotype association in severe sepsis identified by a novel Multi-Individual Array for rapid screening and replication of risk SNPs. Clin Chim Acta. 2012 Jan 18;413(1-2):39-47. doi: 10.1016/j.cca.2011.05.023. Epub 2011 May 25. PMID 21640086
- [Background] Giamarellos-Bourboulis EJ, Netea MG, Rovina N, Akinosoglou K, Antoniadou A, Antonakos N, Damoraki G, Gkavogianni T, Adami ME, Katsaounou P, Ntaganou M, Kyriakopoulou M, Dimopoulos G, Koutsodimitropoulos I, Velissaris D, Koufargyris P, Karageorgos A, Katrini K, Lekakis V, Lupse M, Kotsaki A, Renieris G, Theodoulou D, Panou V, Koukaki E, Koulouris N, Gogos C, Koutsoukou A. Complex Immune Dysregulation in COVID-19 Patients with Severe Respiratory Failure. Cell Host Microbe. 2020 Jun 10;27(6):992-1000.e3. doi: 10.1016/j.chom.2020.04.009. Epub 2020 Apr 21. PMID 32320677
- [Background] Gotts JE, Matthay MA. Endogenous and exogenous cell-based pathways for recovery from acute respiratory distress syndrome. Clin Chest Med. 2014 Dec;35(4):797-809. doi: 10.1016/j.ccm.2014.08.015. Epub 2014 Sep 24. PMID 25453426
- [Background] Haberle H, Magunia H, Lang P, Gloeckner H, Korner A, Koeppen M, Backchoul T, Malek N, Handgretinger R, Rosenberger P, Mirakaj V. Mesenchymal Stem Cell Therapy for Severe COVID-19 ARDS. J Intensive Care Med. 2021 Jun;36(6):681-688. doi: 10.1177/0885066621997365. Epub 2021 Mar 5. PMID 33663244
- [Background] Lai RC, Arslan F, Lee MM, Sze NS, Choo A, Chen TS, Salto-Tellez M, Timmers L, Lee CN, El Oakley RM, Pasterkamp G, de Kleijn DP, Lim SK. Exosome secreted by MSC reduces myocardial ischemia/reperfusion injury. Stem Cell Res. 2010 May;4(3):214-22. doi: 10.1016/j.scr.2009.12.003. Epub 2010 Jan 4. PMID 20138817
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Monsel A, Zhu YG, Gudapati V, Lim H, Lee JW. Mesenchymal stem cell derived secretome and extracellular vesicles for acute lung injury and other inflammatory lung diseases. Expert Opin Biol Ther. 2016 Jul;16(7):859-71. doi: 10.1517/14712598.2016.1170804. Epub 2016 Apr 12. PMID 27011289
- [Background] Shah TG, Predescu D, Predescu S. Mesenchymal stem cells-derived extracellular vesicles in acute respiratory distress syndrome: a review of current literature and potential future treatment options. Clin Transl Med. 2019 Sep 12;8(1):25. doi: 10.1186/s40169-019-0242-9. PMID 31512000
- [Background] Shi Y, Wang Y, Shao C, Huang J, Gan J, Huang X, Bucci E, Piacentini M, Ippolito G, Melino G. COVID-19 infection: the perspectives on immune responses. Cell Death Differ. 2020 May;27(5):1451-1454. doi: 10.1038/s41418-020-0530-3. Epub 2020 Mar 23. No abstract available. PMID 32205856
- [Background] Shi L, Huang H, Lu X, Yan X, Jiang X, Xu R, Wang S, Zhang C, Yuan X, Xu Z, Huang L, Fu JL, Li Y, Zhang Y, Yao WQ, Liu T, Song J, Sun L, Yang F, Zhang X, Zhang B, Shi M, Meng F, Song Y, Yu Y, Wen J, Li Q, Mao Q, Maeurer M, Zumla A, Yao C, Xie WF, Wang FS. Effect of human umbilical cord-derived mesenchymal stem cells on lung damage in severe COVID-19 patients: a randomized, double-blind, placebo-controlled phase 2 trial. Signal Transduct Target Ther. 2021 Feb 10;6(1):58. doi: 10.1038/s41392-021-00488-5. PMID 33568628
- [Background] Shi L, Wang L, Xu R, Zhang C, Xie Y, Liu K, Li T, Hu W, Zhen C, Wang FS. Mesenchymal stem cell therapy for severe COVID-19. Signal Transduct Target Ther. 2021 Sep 8;6(1):339. doi: 10.1038/s41392-021-00754-6. PMID 34497264
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] J. Bindja, M. E. Weiss, M. Schmolz, G. M. Stein, J. Mapes, N. Schneiderhan-Marra, T. O. Joos, E. M. Schneider. Synthetic ligands against TLR2-9 in TruCulture™ - whole blood assays distinguish clinical stages of SIRS (trauma) and sepsis.Trauma, Shock, Inflammation and Sepsis.Trauma, Shock, Inflammation and Sepsis - TSIS 2010; 55 - 63
- [Result] Sanders J., Schneider E.M. How severe RNA virus infections such as SARS-CoV-2 disrupt tissue and organ barriers-Reconstitution by mesenchymal stem cell-derived exosomes. Tissue Barriers in Disease, Injury and Regeneration 2021:95-113. doi: 10.1016/B978-0-12-818561-2.00004-7. Epub 2021 Jun 25. PMCID: PMC8225928.